CLINICAL TRIAL: NCT02393924
Title: UK - A Disease Registry Study to Prospectively Observe Treatment Patterns and Outcomes in Patients With HER2-Positive Unresectable Locally Advanced or Metastatic Breast Cancer
Brief Title: Human Epidermal Growth Factor Receptor 2 (HER2) Positive Unresectable Locally Advanced or Metastatic Breast Cancer Disease Registry Study
Acronym: ESTHER
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML29659
Record Dates: First submitted 2015-03-12; First posted 2015-03-20 (Estimated); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants With HER2-Positive Breast Cancer: Enrolled participants will receive treatment and clinical assessments for their HER2-positive unresectable LABC/mBC as determined by their treating physician, according to the standard of care and routine clinical practice at each site. Participants will be followed until death, withdrawal of consent or study termination, whichever occurs first. Study protocol does not specify any particular drug or treatment regimen.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
This disease registry is a prospective, multicenter non-interventional study designed to observe the different anticancer treatment regimens and their sequencing throughout the course of the disease in participants with unresectable locally advanced breast cancer (LABC) or metastatic breast cancer (mBC) and to describe the clinical outcome for each treatment regimen measured as progression-free survival.

ELIGIBILITY:
Inclusion Criteria:

* Initially diagnosed with HER2-positive unresectable LABC or mBC no more than 6 months prior to enrollment, although they can have received anti-cancer treatment during that time
* Able and willing to provide written informed consent and to comply with the study protocol

Exclusion Criteria:

- There are no exclusion criteria for entry into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with HER2-positive unresectable LABC or mBC
Sampling Method: Probability Sample
Enrollment: 311 (Actual)
Dates: Start 2015-02-23 (Actual); Primary Completion 2023-04-19 (Actual); Study Completion 2023-04-19 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Receiving Each Unique Treatment Regimen Overall | Baseline up to approximately 8 years
Percentage of Participants Receiving Each Unique Treatment Regimen as First-Line Versus Subsequent-Line Therapy | Baseline up to approximately 8 years
Percentage of Participants Receiving Each Unique Treatment Regimen Sequence | Baseline up to approximately 8 years
Progression-Free Survival | From start date of anti-cancer treatment regimen to the date of either disease progression or death (up to approximately 8 years)
  Tumor response will be evaluated by the Investigator according to site-specific medical practice. Study protocol does not specify any particular method of assessment.

SECONDARY OUTCOMES:
Overall Survival (OS) | From the date of initiation of treatment to the date of death from any cause (up to approximately 8 years)
Percentage of Participants With Objective Response of Complete Response (CR) or Partial Response (PR) | From the date of initiation of treatment to the date of disease progression or death from any cause (up to approximately 8 years)
  Tumor response will be evaluated by the Investigator according to site-specific medical practice. Study protocol does not specify any particular method of assessment.
Duration of Response (DoR) | From date of first response (CR or PR) to the date of disease progression (up to approximately 8 years)
  Tumor response will be evaluated by the Investigator according to site-specific medical practice. Study protocol does not specify any particular method of assessment.
Time to Treatment Failure | From the date of initiation of treatment to the date of treatment stopped or switched or death from any cause (up to approximately 8 years)
Percentage of Participants With Central Nervous System (CNS) as First Site of Progression | From the date of initiation of treatment to the date of disease progression or death from any cause (up to approximately 8 years)
Percentage of Participants With Adverse Events (AEs) and Serious AEs (SAEs) | Baseline up to approximately 8 years
Percentage of Participants by Reasons for Treatment Modification | Baseline up to approximately 8 years
Percentage of Participants Receiving Each Treatment Regimen Categorized by Participant Characteristics | Baseline up to approximately 8 years
Number of Treatment Regimens Received | Baseline up to approximately 8 years
Euro Quality of Life 5-Dimension Questionnaire (EQ-5D) Score | Baseline up to approximately 8 years (assessed every 3 months)
Functional Assessment of Cancer Therapy-Breast (FACT-B) Questionnaire Score | Baseline up to approximately 8 years (assessed every 3 months)
Work Productivity and Activity Impairment (WPAI) Questionnaire Score | Baseline up to approximately 8 years (assessed every 3 months)
Percentage of Participants with Different Anti-Cancer Treatment Regimens by Country | Baseline up to approximately 8 years
Percentage of Participants with History of Breast Cancer by Different Anti-Cancer Treatment Regimens | Baseline up to approximately 8 years
Percentage of Participants with CNS-only Disease Progression | From the date of initiation of treatment to the date of disease progression or death from any cause (up to approximately 8 years)
Percentage of Participants with Oligometastatic Disease Categorized by Different Anti-Cancer Treatment Regimens | Baseline up to approximately 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (30):
- United Kingdom (30):
  - Kent & Canterbury Hospital, Canterbury
  - Chesterfield Royal Hospital, Chesterfield
  - Royal Cornwall Hospital; Dept of Clinical Oncology, Cornwall
  - Castle Hill Hospital; The Queens Centre for Oncology and Haematology, Cottingham
  - Hairmyres Hospital; Oncology Dept, East Kilbride
  - Queen Elizabeth Hospital, Gateshead
  - Raigmore Hospital, Inverness
  - Forth Valley Royal Hospital ; Oncology Department, Larbert
  - Queen Elizabeth Hospital, London
  - Royal Marsden Hospital; Dept of Med-Onc, London
  - Charing Cross Hospital; Medical Oncology., London
  - Macclesfield District General Hospital, Macclesfield
  - Maidstone Hospital; Kent Oncology Centre, Maidstone
  - Christie Hospital Nhs Trust; Medical Oncology, Manchester
  - James Cook University Hospital; Oncology and Radiology, Middlesbrough
  - Northampton General Hospital NHS Trust;Oncology Unit, Northampton
  - Mount Vernon & Watford Trust Hospital; Dept. of Clinical Oncology, Northwood
  - Norfolk & Norwich University Hospital; Oncology Department, Norwich
  - Nottingham City Hospital; Oncology, Nottingham
  - Derriford Hospital; Plymouth Oncology Centre, Plymouth
  - Royal Preston Hosp; Rosemere Cancer Ctr, Preston
  - North Wales Cancer Treatment Centre, Glan Clwyd Hospital, Rhyl
  - Scarborough General Hospital, Scarborough
  - Royal Shrewsbury Hospitals Nhs Trust; Oncology, Shrewsbury
  - Royal Marsden Hospital; Dept of Medical Oncology, Sutton
  - Singleton Hospital; Pharmacy, Swansea
  - Great Western Hospital, Swindon Cancer Research Unit; Osprey Unit Level 3, Swindon
  - Pinderfields Hospital; Clinical Research Team, Rowan House, Wakefield
  - Yeovil District Hospital; Macmillan Unit, Yeovil
  - Airedale General Hospital; Oncology, York

REFERENCES:
- [Derived] Ring A, Sutherland S, Harper-Wynne C, Owen J, Sanglier T, Velikova G. A disease registry study to prospectively observe treatment patterns and outcomes in patients with HER2-positive unresectable LA/MBC: final results of the ESTHER study. Breast Cancer Res Treat. 2025 Jul;212(1):113-121. doi: 10.1007/s10549-025-07708-4. Epub 2025 May 13. PMID 40358647